CLINICAL TRIAL: NCT07364786
Title: Intratumoral Pressure, Intratumoral Partial Oxygen Pressure, and Inflammatory Cytokines in Antisecretory Factor Treatment of Glioblastoma
Brief Title: Effect of Salovum® on Pressure, Oxygen and Inflammation in Glioblastoma
Acronym: AFGBMBiop
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Siesjö (Other)
Collaborators: Lund University (Other); Region Skane (Other)
Responsible Party: Sponsor-Investigator, Peter Siesjö, MD, PhD, Consultant Neurosurgeon, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AFGBMBiopsi.v7
Record Dates: First submitted 2024-10-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; interstitial fluid pressure; cytokine; diagnostic biopsy; partial oxygen pressure; antisecretory factor
MeSH Terms: conditions — Glioblastoma | interventions — antisecretory factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salovum (Experimental): Ingestion of Salovum during 48 hours starting 24 hours after diagnostic biopsy
  Interventions: Dietary Supplement: Salovum

INTERVENTIONS:
Dietary Supplement: Salovum — Ingestion of Salovum 11g three times daily during 48 hours
  Other Names: Antisecretory factor

SUMMARY:
The objective of this clinical trial is to investigate the effects of Salovum®, an egg yolk powder enriched with the endogenous protein antisecretory factor, in participants undergoing diagnostic biopsies for suspected glioblastoma. The primary questions the trial seeks to answer are:

* Will Salovum® reduce intratumoral pressure?
* Will Salovum® influence the release of inflammatory cytokines from tumor tissue? Additionally, the study will investigate the impact of Salovum® on intratumoral partial oxygen pressure and tumor volume.

Researchers will:

* Place probes for measuring intratumoral pressure, microdialysis, and partial oxygen pressure during a standard biopsy procedure.
* Compare measurements from participants before and during ingestion of Salovum®.

Participants will:

* Have probes implanted during a surgical biopsy.
* Ingest Salovum® 24 to 72 hours after the procedure.

DETAILED DESCRIPTION:
Background and Rationale Glioblastoma is the most prevalent primary brain tumor and has the poorest prognosis. Antisecretory factor (AF) is a crucial 41 kDa endogenous protein initially identified for its ability to inhibit experimental diarrhea. The active amino-terminal segment of AF has been synthesized into a 16-amino acid peptide (AF-16) and utilized in animal studies. Salovum®, a product based on the egg yolk powder B221®, contains high levels of AF and is classified as a "food for special medical purposes" by the European Food Safety Agency. It is available over-the-counter in Swedish pharmacies. Specially processed cereals (SPC®) have been shown to induce circulating AF after ingestion.

Many tumors, including glioblastoma, exhibit higher interstitial fluid pressure (IFP) than surrounding tissues, potentially hindering chemotherapy penetration in systemic treatments and possibly increasing excretion during intratumoral treatments.

In head injury models, AF has been effective in reducing elevated intracranial pressure and improving functional outcomes. Similarly, AF has demonstrated a significant reduction in intracranial pressure and increased survival rates in an experimental model of herpes encephalitis. Preliminary results from our studies indicate that treatment with antisecretory factor in patients with severe traumatic head injuries reduces intracranial pressure and improves treatment outcomes. Since Salovum® is not classified as a drug, clinical trials have only required ethics approval.

AF is an endogenous protein, and no antibody formation has been observed when administered to humans. Despite being administered to hundreds of patients, no side effects have been reported. Egg yolk allergy is a contraindication, though no cases of triggered allergies have been documented. In mouse models of malignant brain tumors, AF-16, Salovum® , or SPC® have been shown to lower interstitial fluid pressure and enhance the efficacy of both systemic and intratumoral temozolomide treatment. AF-16 also exhibits immunomodulatory effects on myeloid cells in vitro and on the secretion of immunomodulatory substances from tumor cells. It remains unclear whether AF's effects in tumor models are due to its antisecretory or immunomodulatory properties, or if the former is a result of the latter. Modulation of circulating complement complexes with proteasome units has also been suggested as a potential mechanism.

Details of Trial Diagnostic biopsies will be performed according to clinical routine under general anesthesia, using intraoperative navigation. Subsequently, two intracranial pressure sensors and one microdialysis catheter (for the first five patients) will be inserted through the same burr hole. One pressure sensor and the microdialysis catheter will be placed inside the tumor tissue, and another pressure sensor will be placed outside the tumor tissue. For the next five patients, an oxygen sensor and a microdialysis catheter will be placed inside the tumor tissue, and an oxygen sensor outside the tumor tissue. The catheters will be fixed in a bone-anchored four-lumen bolt.

In both groups, pressure and partial oxygen pressure will be recorded for approximately 24 hours, followed by the administration of Salovum as described above, with sampling continuing for 48 hours. The catheters will then be removed bedside after local anesthetics. Pressure will be recorded using input pressure sensors (Pressio® ICP, Sophysa), with data stored in dedicated hardware and software (Pressio monitoring system, Sophysa). Partial oxygen pressure will be continuously recorded using a CNS monitor (Moberg ICU solutions), and microdialysis will be conducted with CMA 100 catheters and existing hardware and software. The insertion of pressure sensors, oxygen sensors, and microdialysis catheters is standard clinical practice in the treatment of head injuries and subarachnoid hemorrhages.

The risk of bleeding and infection requiring treatment in diagnostic brain tumor biopsy is below 1%. The insertion of catheters as described is not expected to present a measurable additional risk of bleeding and/or infection. In previous cases where we inserted two microdialysis catheters in eight patients with glioblastoma, no side effects such as bleeding or infection were recorded. The described catheter insertion procedure is estimated to extend the operation time by about 20 minutes.

Ethical Considerations Glioblastoma carries a grim prognosis. Antisecretory factor has shown promising results in combination with chemotherapy in experimental models of human and mouse brain tumors. A clinical open phase 2 trial has demonstrated the safety and feasibility of this treatment, with no reported side effects from Salovum®. As with all studies involving serious and fatal diseases, there is an ethical consideration regarding the hope for treatment efficacy. Both oral and written information will emphasize that there are no guarantees of treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected glioblastoma
2. Age 18-75 years
3. Planned diagnostic biopsy
4. Informed consent of subject

Exclusion Criteria:

1. Known egg yolk allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Intratumoral pressure after ingestion of Salovum® | 0 to 72 hours after diagnostic biopsy
  To measure intratumoral pressure by insertion of catheters to measure pressure (Sophysa, France) before and during ingestion of Salovum® in participants diagnosed with glioblastoma (GBM) who undergo a diagnostic biopsy.

SECONDARY OUTCOMES:
Inflammatory cytokine release after ingestion of Salovum® | 0 to 72 hours after diagnostic biopsy
  To measure inflammatory cytokine release by sampling of extracellular fluid with a microdialysis probe (Dialysis, Sweden) and analysis by multiplex arrays (Mesoscale Discovery, US) before and during ingestion of Salovum® in participants diagnosed with glioblastoma (GBM) who undergo a diagnostic biopsy.

OTHER OUTCOMES:
Intratumoral partial oxygen pressure after ingestion of Salovum® | 0 to 72 hours after diagnostic biopsy
  To measure intratumoral partial oxygen pressure by inserted catheters and monitor (LICOX, US) before and during ingestion of Salovum® in participants diagnosed with glioblastoma (GBM) who undergo a diagnostic biopsy.
Tumor volume after ingestion of Salovum® | At time of standard follow up MRI 3-4 months after a diagnostic biopsy
  To measure tumor volume in participants given Salovum® after a diagnostic biopsy for suspected glioblastoma
Intratumoral pressure versus intracerebral pressure | 0-72 hours
  To measure the difference in intratumoral and intracerebral pressure by insertion of catheters to measure pressure (Sophysa, France) before and after ingestion of Salovum® in participants who undergo a diagnostic biopsy for suspected glioblastoma
Intratumoral partial oxygen pressure versus intracerebral partial oxygen pressure | 0-72 hours
  To measure the difference in intratumoral and intracerebral partial oxygen pressure by inserted catheters and monitor (LICOX, US) before and after ingestion of Salovum® in participants who undergo a diagnostic biopsy for suspected glioblastoma

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siesjö, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Department of Neurosurgery, Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided